CLINICAL TRIAL: NCT01245569
Title: A 12-week, Multicentre, Multinational, Randomized, Double-blind, Double-dummy, 2-arm Parallel Group Study Comparing the Efficacy and Safety of Foster® 100/6 (Beclomethasone Dipropionate 100 µg Plus Formoterol 6 µg/Actuation), 2 Puffs b.i.d., Versus Seretide® 500/50 (Fluticasone 500 µg Plus Salmeterol 50 µg/Actuation), 1 Inhalation b.i.d., in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study in Patients With Chronic Obstructive Pulmonary Disease
Acronym: FUTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0910-PR-0021; 2009-014410-10 (EudraCT Number)
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foster® (Experimental): Foster® (beclomethasone dipropionate 100 µg plus formoterol 6 µg/unit dose), 2 inhalations b.i.d. (daily dose of BDP "extrafine" 400 µg plus FF 24 µg).
  Interventions: Drug: Foster® 100/6 µg/unit dose
- Seretide® Accuhaler® (Active Comparator): Seretide® Accuhaler® (fluticasone 500 μg plus salmeterol 50 μg/actuation), 1 inhalation b.i.d. (daily dose of fluticasone 1000 μg plus salmeterol 100 μg).
  Interventions: Drug: Seretide Accuhaler® 500/50 µg/actuation

INTERVENTIONS:
Drug: Foster® 100/6 µg/unit dose — Foster® (beclomethasone dipropionate 100 µg plus formoterol 6 µg/unit dose), 2 inhalations b.i.d. (daily dose of BDP "extrafine" 400 µg plus FF 24 µg).
  Arms: Foster®
Drug: Seretide Accuhaler® 500/50 µg/actuation — Seretide® Accuhaler® (fluticasone 500 μg plus salmeterol 50 μg/actuation), 1 inhalation b.i.d. (daily dose of fluticasone 1000 μg plus salmeterol 100 μg).
  Arms: Seretide® Accuhaler®

SUMMARY:
The purpose of the present study is to determine the effects on health status and spirometric values of Foster® 100/6 (two puffs b.i.d.) versus Seretide® 500/50 (one inhalation b.i.d.), over a 12-week treatment period in Chronic Obstructive Pulmonary Disease (COPD) patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is an incurable, debilitating and progressive disease that can be fatal. The recent Global Burden of Disease Study ranks COPD as the 6th leading cause of mortality and the 12th leading cause of morbidity world-wide. Furthermore, trends in the use of medical care resources indicate that the economic cost of COPD continues to rise in direct relation to the ageing population, the increase in prevalence of disease and the cost of new and existing medical and public health interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 40 years, who have signed an Informed Consent form prior to initiation of any study-related procedure or once applicable written informed consent obtained by legal representative.
2. Outpatients with a diagnosis of COPD and including:

   1. Smoking history of at least 10 pack years defined as [(number of cigarettes smoked per day) x (number of years of smoking) / 20], both current and ex-smokers are eligible.
   2. Use of bronchodilators in the previous 2 months to visit 1.
   3. Post-bronchodilator FEV1 < 60% of the predicted normal value.
   4. Post-bronchodilator FEV1/FVC < 0.7.
   5. A ≥ 5% response to a reversibility test.
   6. A Baseline Dyspnoea Index (BDI) focal score less or equal than 10 (to be met also at visit 2).
3. History of no more than one COPD exacerbation in the previous 12 months (without considering the last 2 months) to visit 1.
4. A cooperative attitude and ability to be trained to the proper use of pMDI and DPI (Accuhaler®, circular moulded plastic inhaler) inhalers.

Main Exclusion Criteria:

1. Clinically relevant respiratory disorders.
2. Current diagnosis of asthma or respiratory disorders other than COPD.
3. Clinically significant laboratory and ECG abnormalities indicating a significant or unstable concomitant disease which may impact the feasibility of the results of the study according to investigator's judgement.
4. Patients with COPD exacerbation in the 2 months prior to screening and during the study period.
5. Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia.
6. Patients treated with depot corticosteroids in the 2 months preceding the visit 1 and during the run-in period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Transition Dyspnoea Index (TDI) score | At day 84
Area Under the Curve (AUC) 0-30min standardized by time of change from pre-dose in Forced Expiratory Volume in one second (FEV1) | After drug inhalation in the morning of day 1

SECONDARY OUTCOMES:
Change from baseline in pre-dose morning Forced Expiratory Volume in one second (FEV1) | At each clinic visit
Change from pre-dose in Forced Vital Capacity (FVC) | At 5, 15, 30 min after drug intake, at day 1 and day 84
Change from baseline in the St George's Respiratory Questionnaire (SGRQ)component and total scores | At day 84
Change from baseline in pre-dose and in post-dose distance walked (6 Minute Walking Test - 6MWT) (in a subset of at least 50 % of patients from pre-selected sites) | At day 84

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — The Medicine Evaluation Unit - Manchester, UK; Jorgen Vestbo, MD, Principal Investigator — Dept. of Cardiology and Respiratory Medicine - Copenhagen, Denmark
Locations (1):
- Policlinico Umberto I - VIII Padiglione, Rome, Rome, Italy

REFERENCES:
- [Result] Singh D, Nicolini G, Bindi E, Corradi M, Guastalla D, Kampschulte J, Pierzchala W, Sayiner A, Szilasi M, Terzano C, Vestbo J; FUTURE (Foster Upgrades TherapeUtic care in REspiratory disease) study group. Extrafine beclomethasone/formoterol compared to fluticasone/salmeterol combination therapy in COPD. BMC Pulm Med. 2014 Mar 12;14:43. doi: 10.1186/1471-2466-14-43. PMID 24621109
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2009-014410-10